CLINICAL TRIAL: NCT00256373
Title: Treatment of Chronic Low Back Pain: A Trial Comparing Traditional Back School and Individual Therapist-Assisted Exercise
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Collaborators: Sygekassernes Helsefond (Other); Apotekerfonden af 1991 (Other); Indenrigs- og sundhedsministeriet (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KA 01011
Record Dates: First submitted 2005-11-16; First posted 2005-11-21 (Estimated); Last update posted 2006-04-19 (Estimated); Status verified 2005-09

CONDITIONS: Chronic Low Back Pain
Keywords: Low Back Pain; Dynamic Back-Muscle exercise Treatment; Interdisciplinary Treatment; Roland Morris Disability Questionnaire; SF-36; Low Back Pain Rating Scale
MeSH Terms: conditions — Low Back Pain

INTERVENTIONS:
Procedure: Mod. functional restoration-Individ. dynamic back-muscle

SUMMARY:
Rheumatologists are discussing, whether rehabilitation of patients with low back pain (LBP) can be improved. At present patients with LBP start treatment as soon as possible, this also applies for patients with chronic low back pain (CLBP) - pain lasting over 12 weeks. At Glostrup University Hospital department of Physical Medicine/rheumatology we use a method (method A) where an interdisciplinary team gives the patients a treatment composed of various topics. This includes among other things education, physical team training, exercises in swimming pool, stretching exercises, and occupational therapy. A different method (method B) originates from the Rehabilitation centre in Karlslunde led by Teddy Oefeldt. Here they focus strictly on dynamic training of muscles in the back and the buttocks. A therapist, who in the beginning partly carries the patient through the exercises, assists this training.

In both methods, individually considerations are taken, but to a greater extend in method B. The treatment will extend over a three months period.

A few earlier investigations have compared these two methods, but they have not been systematized to such a degree, that they gave any final conclusions. Therefore, we initialized an investigation including a larger number of patients, where the two methods are compared from the results the patients achieve after 3, 6, 12 and 24 months.

286 consecutive patients were included and randomized to one of the two methods. Those, who did not wish to participate in the investigation, were treated according to the department's normal procedure (Method A)

ELIGIBILITY:
Inclusion Criteria:

1. Low Back Pain lasting more than 12 weeks with or with out pain radiating into the leg(s)
2. Age 18 - 60 years

Exclusion Criteria:

1. Serious spinal pathology

   1. Malignancy
   2. Osteoporosis,
   3. Fresh vertebral fracture
   4. Newly operation on the back
   5. Stenosis of the lumbar spine
   6. Unstable spondylolistesis
   7. Infections in the back
2. Neurological dysfunction of the thoracic or abdominal muscles
3. Pregnancy/breastfeeding
4. Mental illness
5. Health conditions which prohibit intensive training.
6. Languish problems/ dyslexia

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2001-01; Study Completion 2005-11

PRIMARY OUTCOMES:
Pain VAS

SECONDARY OUTCOMES:
Roland Morris Disability Questionnaire
SF-36
Low Back Pain Rating Scale
Medicine use
Work situation
Pension
Change in physical activity
Global assessment

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Lundsgaard, MD, Study Chair; Claus Hellesen, MD, Study Director; Alex Oefeldt, Therapist, Study Director; Gorm Thamsborg, Dr.Med.Sci., Study Director; Arne Astrup, Dr.Med.Sci., Study Director; Steen Stender, Dr.Med.Sci., Study Chair; Ninna Dufour, MD, Principal Investigator — Unfilliated
Locations (1):
- Glostrup University Hospital, Glostrup Municipality, Denmark

REFERENCES:
- [Derived] Dufour N, Thamsborg G, Oefeldt A, Lundsgaard C, Stender S. Treatment of chronic low back pain: a randomized, clinical trial comparing group-based multidisciplinary biopsychosocial rehabilitation and intensive individual therapist-assisted back muscle strengthening exercises. Spine (Phila Pa 1976). 2010 Mar 1;35(5):469-76. doi: 10.1097/BRS.0b013e3181b8db2e. PMID 20147878